CLINICAL TRIAL: NCT03529032
Title: A Preoperative Methadone Single Dose for Moderately to Severely Painful Surgery Reduces Postoperative Morphine Consumption Results From a Double-blind Pragmatic Clinical Trial
Brief Title: Preoperative Methadone Single Dose Reduces Postoperative Morphine Consumption.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kantonsspital Baden (Other)
Responsible Party: Principal Investigator, Philipp Bühler, MD, MD, Kantonsspital Baden
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ref.Nr.EK:2011/052
Record Dates: First submitted 2013-07-12; First posted 2018-05-18 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Pain, Postoperative
Keywords: methadone; postoperative pain; acute pain therapy; postoperative pain therapy
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl group (No Intervention): Drug: Fentanyl Fentanyl group 3µg/kg to start surgery TIVA: general anesthesia will be based on Fentanyl an Propofol, titrated to achieve bispectral index (BIS) between 40-60.
- methadone group (Experimental): Drug: methadone methadone group 0.2mg/kg to start surgery TIVA: general anesthesia will be based on Fentanyl an Propofol, titrated to achieve bispectral index (BIS) between 40-60.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — methadone for control postoperative pain
  Arms: methadone group

SUMMARY:
The aim of this study was to evaluate the effect of intraoperative methadone on postoperative analgesic requirements, pain scores and patient satisfaction in comparison to standard intraoperative pain control with fentanyl.

DETAILED DESCRIPTION:
Patients of both genders and up to age 75 and ASA classification III were enrolled, when undergoing moderately to severely painful surgery scheduled for ≥90 minutes in general anaesthesia. Patients were randomized to receive either a single shot of methadone (0.2mg/kg) or fentanyl (0.003mg/kg) for induction of anesthesia. In cases of insufficient intraoperative analgesia repeated fentanyl administration was possible. Postoperative analgesia was provided with patient controlled morphine in both groups (PCA = Patient Controlled Analgesia). Pain was assessed using the numerical rating scale (NRS) at rest and after coughing, at 15 minutes post extubation, and repeated every 6 hours up to 72 hours postoperatively. The levels of sedation and nausea/vomiting were also evaluated in parallel.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* Patients of both genders and up to age 75 and ASA classification III were enrolled, when undergoing moderately to severely painful surgery scheduled for ≥90 minutes in general anaesthesia.
* german speaking patients

Exclusion Criteria:

* patients including other studies
* pregnant
* breast feeding
* patients in methadone substitution therapy
* dependent drug user
* patients with BMI greater than 36kg/m2
* patients with chronic or acute renal failure with serum creatinine greater than 400µmol/L
* patients with liver insufficiency or failure
* alcoholics
* patients with acute heard attack

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Difference of postoperative morphine consumption | first 48 hours postoperatively
  Difference in milligrams of morphine used as rescue by patient controlled analgesia pump

SECONDARY OUTCOMES:
Difference in pain scores, using the Numeric Rating Scale | first 72 hours postoperatively
  Difference in pain scores in rest and motion at 0,6,12,24,36,48,72 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Buehler, MD, Principal Investigator — Kantonsspital Baden
Locations (1):
- Kantonsspital Baden, Baden, Canton of Aargau, Switzerland